CLINICAL TRIAL: NCT05391802
Title: A Multicenter, Prospective, Single-arm Objective Performance Criteria Trial to Evaluate the Safety and Efficacy of the Transcatheter Mitral Valve Repair System: ValveClasp® in the Treatment of Moderate to Severe Mitral Regurgitation
Brief Title: The Multicenter Clinical Trial of a Novel TEER Decive (V-CLASP Trial)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYYL2022-02ZC-01
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Patients with PMR erolled in the trail will receive transcatheter mitral valve repair using the ValveClasp system
  Interventions: Device: Transcatheter mitral valve repair

INTERVENTIONS:
Device: Transcatheter mitral valve repair — Transcatheter mitral valve repair (TMVr) is a minimally invasive procedure. Doctors place a thin tube (calleda catheter) into a large vein to reach your heart. A clip is then placed onto the center of your mitral valve. The valve continues to open and close, allowing blood to flow through while reducing MR.

SUMMARY:
This is a single-group, prospective, multicenter clinical research using the single-arm objective performance criteria. Patients with moderate to severe mitral regurgitation and a high surgical risk will be treated with ValveClasp®, a novel transcatheter mitral edge-to-edge repair system.

The subjects will be followed postoperatively, before discharge, for one month, six months, and twelve months. immediately following operation, before discharge, and at 1, 6, and 12 months after surgery, with follow-up at 2, 3, 4, and 5 years. The follow-ups began immediately before discharge and continued for one month, six months, and twelve months after surgery, with extensions to two, three, four, and five years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥70 years old.
2. The existence of primary mitral regurgitation of moderate to severe severity or more was established by transthoracic echocardiogram (TTE) or transesophageal echocardiography (TEE) within 3 months previous to inclusion.
3. NYHA class II-IV, symptomatic subject.
4. The subject's left ventricular ejection fraction (LVEF) was less than 20% within the three months preceding to enrolment, as determined by any of the following methods: echocardiography, left ventriculography, or cardiac magnetic resonance imaging (MRI) (not visual assessment).
5. Subjects were evaluated for cardiac anatomical fitness for mitral valve repair surgery as well as suitability for the research device.
6. Subjects were evaluated for femoral access appropriateness and atrial septal puncture feasibility.
7. Patients who have been assessed as having a high or very high surgical risk by the cardiac specialists at each clinical trial location. The most important factor in their decision *Score from the American Association for Thoracic Surgery (STS): 8% for surgical mitral valve replacement and 8% for surgical mitral valve repair.

   STS score of 8% for surgical mitral valve replacement or 6% for surgical mitral valve repair, or the presence of additional surgical high-risk variables (such as** significant weakness or the presence of two or more patients).

   severe frailty, more than two uncorrectable organ failures, and surgical-related impairments (history of open heart surgery, extremely severe thoracic deformity, and so on), with STS ratings based on the website version accessible at the time of registration.

   **According to the 2020 AHA/ACC Guidelines for Valve Management, high risk for mitral valve surgery is defined by FDA and MVARC criteria.
8. The patient is willing and capable of adhering to the protocol's requirements and data collecting methods, understands the trial's aim, and freely participates in and signs the clinical study by himself or a legal guardian. (8) The participant consents willingly and signs a written informed consent form authorized by the Clinical Trial Ethics Committee.

Exclusion Criteria:

1. After heart transplantation, mitral valve surgery or mitral valve transcatheter surgery
2. Acute myocardial infarction within 1 month.
3. Any vascular intervention or surgical procedure within 1 month.
4. The investigator determines that the subject's femoral vein cannot accommodate the largest size catheter in the test product or an ipsilateral deep vein thrombosis.
5. The subject has a medical condition that would make evaluation of treatment difficult (e.g., cancer, infection, severe metabolic disease, severe neurological

(5) Have a disease that would make evaluation of treatment difficult (e.g., cancer, infection, severe metabolic disease, severe neurological lesions affecting cognitive ability, psychiatric disease, etc.); or special cases that have been evaluated by the local trial center cardiac team as inappropriate for (4) Surgical studies related to this clinical trial device. (6) Severe non-mitral valve disease requiring urgent management and other cardiac surgical procedures.

(7) Severe mitral valve calcification; leaflet anatomy not conducive to mitral valve clip placement.

(8) Severe pulmonary hypertension (pulmonary artery systolic pressure >90 mmHg as measured by echocardiography).

(9) Untreated controlled acute pulmonary edema. (10) Severe right heart insufficiency. (11) Bleeding disorders or disorders of coagulation; or the presence of contraindications to antithrombotic therapy (12) Active infection requiring current antibiotic therapy (in the case of transient disease, the patient will not be enrolled until at least 14 days after discontinuation of antibiotics).

(12) Active infection requiring current antibiotic therapy (in the case of temporary disease, patients should be off antibiotics for at least 14 days before being enrolled). Patients must be free of infection prior to treatment and required dental treatment should be completed at least 21 days prior to treatment.

(13) History of acute peptic ulcer or gastrointestinal bleeding within 2 months.

(14) Untreated severe coronary artery stenosis requiring hemodialysis (15) Ultrasound showing intracardiac thrombus, bulky mass, or mass. (16) History of infective endocarditis, rheumatic heart disease. (17) Hemodynamic instability, defined as systolic blood pressure <90 mmHg without afterload-reducing drugs, uncorrected cardiogenic shock or the use of intra-aortic balloon counterpulsation. (18) Patients with contraindications to transesophageal echocardiography (TEE) and contraindications to general anesthesia.

(19) Patients with allergies or contraindications to study devices or surgical drugs that cannot be adequately managed by medical means (20) Life expectancy <12 months due to concomitant non-cardiac comorbidities. (21) Subjects are participating in other clinical trials that have not met the observed endpoints or that would clinically interfere with this clinical trial (21) An experimental drug or other device study in which the subject is participating in another clinical trial that has not met the observed endpoint or would clinically interfere with the study endpoint of this clinical trial. (Note: If a trial requires extended follow-up of a product that was investigational at the time of the trial but has since been marketed, the trial should be conducted in a manner that is consistent with the clinical trial. (Note: If a trial requires extended follow-up of a product that was investigational at the time of the trial but has since been marketed, the trial is not considered to be an investigational trial).

(22) Patients who, in the opinion of the investigator, are not suitable for enrollment in this trial.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Treatment efficiency rate | 0-360 days
  Treatment efficiency defined as no death, no incidence of mitral valve reoperation, MR ≤2+) at 12 months postoperatively.

SECONDARY OUTCOMES:
Operation success rate | 0-360 days
  Operation success defined as Successful device delivery, release, and implantation; implanted mitral valve clamps in the correct position; and implanted mitral valve clamps attaining the targeted efficacy (mitral regurgitation 2+ and mean transvalvular pressure difference 5 mmHg)

IPD SHARING:
Plan to Share IPD: No